CLINICAL TRIAL: NCT05406011
Title: Effect of Sour Cherry Anthocyanins (Cyanidin Components of Sour Cherry) on Human Saliva and Biofilm Formation
Brief Title: Effect of Sour Cherry Anthocyanins on Healthy Human Saliva
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Debrecen (Other)
Responsible Party: Principal Investigator, Dr. Boglárka Emese Skopkó, Department of Dentoalveolar Surgery, assistant lecturer, University of Debrecen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-IV/1120-1/2020
Record Dates: First submitted 2022-03-11; First posted 2022-06-06 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Anthocyanins; Tooth Exfoliation

STUDY DESIGN:
Intervention Model Description: The participants are subdivided in parallel groups by their age and according to the toothbrush change (to change or not to change the toothbrush) after scaling.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Age groups (Experimental): Participants grouped by their age (Age group I: patients aged between 18-30, age group II: patients aged between 31-45).
  Interventions: Dietary Supplement: Pelleted sour cherry (anthocyanin) containing chewing gum usage.; Dietary Supplement: Pelleted chewing gum for stimulated saliva sampling.; Procedure: Scaling
- Groups by toothbrush change (Experimental): Half of the group change the toothbrush after scaling and the other half not.
  Interventions: Dietary Supplement: Pelleted sour cherry (anthocyanin) containing chewing gum usage.; Dietary Supplement: Pelleted chewing gum for stimulated saliva sampling.; Procedure: Scaling
- Experimental period (Experimental): Control: Control period without sour cherry chewing gum usage, with saliva sampling on fixed appointments (between 12:00 and 14:00, 0th, 4th and 7th day of the week) of the week. At the beginning oral and basic periodontal examinations performed. Plaque and calculus index at every sampling occasions.
  Prevention: After a full mouth scaling sour cherry chewing gum usage, for a week. Saliva sampling on the same days. Plaque and calculus index at every sampling occasions.
  Therapeutic: Sour cherry chewing gum usage, for one more week. Saliva sampling on the same days. Plaque and calculus index at every sampling occasions.
  Control (without sour cherry chewing gum usage), prevention and therapeutic periods takes 3 weeks together.
  Interventions: Dietary Supplement: Pelleted sour cherry (anthocyanin) containing chewing gum usage.; Dietary Supplement: Pelleted chewing gum for stimulated saliva sampling.; Procedure: Scaling

INTERVENTIONS:
Dietary Supplement: Pelleted sour cherry (anthocyanin) containing chewing gum usage. — Dietary Supplement usage (daily 3 times for 2 weeks) with salivary sampling on fixed days (1., 4. and 7.) and daytime (between 12:00 and 14:00) of the week. Procedure: Scaling after a control period without sour cherry chewing gum usage (1 week).
Dietary Supplement: Pelleted chewing gum for stimulated saliva sampling. — Stimulated saliva sampling after chewing a pelleted gum without active ingredient (used only before stimulated saliva sampling), during the whole experimental period (control and parallel with sour cherry chewing gum usage) with sampling on fixed days (1., 4. and 7.) and daytime (between 12:00 and 14:00) of the week.
Procedure: Scaling — Scaling after a 1-week control period without chewing the sour cherry gum.

SUMMARY:
The experiment is based on earlier research where it was proven that chewing gum usage with anthocyanin rich sour cherry extract significantly reduces the amount of human salivary alpha-amylase in unstimulated saliva samples and stimulated saliva samples taken in every 10 minutes till a half an hour as compared to placebo. The S. mutans counts' number on agar base cultures were greater in case of the stimulated samples of placebo and anthocyanin containing chewing gum groups.

The investigators' aims were to extend the background of the earlier established phenomena: The sour cherry (anthocyanin) containing chewing gum usage (around 2 weeks, daily 3 times) is beneficent on the human oral microflora and cytokine level/expression.

DETAILED DESCRIPTION:
The experiment is based on earlier research where it was proven that chewing gum usage with anthocyanin rich sour cherry extract significantly reduces the amount of human salivary alpha-amylase in unstimulated saliva samples and stimulated saliva samples taken in every 5 minutes till a half an hour as compared to placebo.

The investigators' study: Examination the effect of sour cherry anthocyanin containing chewing gum in a study taking a 3-week experimental period. At the beginning of experimental period oral and basic periodontal examination of the participants. Selection of healthy young adults (10 person) and adults (10 person), who has good oral hygiene, do not suffer from serious general disease and do not get respiratory infection treated with antibiotics in the past 2 months. Arranging saliva sampling on fixed appointments (between 12:00 and 14:00, 1st, 4th and 7th day of the week) through 3 weeks. On the 1. week, which is a control period taking of resting saliva samples and stimulated saliva samples from the participants. The stimulated saliva sampling is made after chewing of a gum without active ingredient. At the end of the control week a full mouth scaling is made and after it all of the participants get sour cherry containing chewing gums to chew 3x daily till 2 weeks, and the sampling occasions arranged on the same days as on the control week. After scaling 10 participant change their toothbrush, and 10 do not change. The saliva sample analyzation is placed in the Institute of Food Technology, the Department of Human Genetics and Department of Microbiology where they are frozen on -80 Celsius till the laboratory analysis.

16S (16 Svedberg) rRNA (ribosomal ribonucleic acid) sequencing is starting with DNA isolation by Inhibitor Removal Technology followed by sequencing with Illumina MiSeqSystem. PCR (Polymerase Chain Reaction) analysis of saliva samples starting with RNA isolation of samples with MagMAX Viral Kit, followed by RNA transcription and qPCR (quantitative polymerase chain reaction ) according to the Manufacturer's Instructions. ELISA (Enzyme Linked Immunosorbent Assay) analysis with appropriate saliva analyzation kit for the listed cytokines as follows: Examined cytokines (PCR and ELISA): Interleukins: Interleukin-1β, Interleukin-2, Interleukin-6; TNF(tumor necrosis factor) alfa, Melatonin (ELISA) , Mucin 7 (ELISA) and Mucin-5B (5subtypeB) (ELISA).

The investigators' aims to are to extend the background of the earlier established phenomena: The sour cherry (anthocyanin) containing chewing gum usage (around 2 weeks, daily 3 times) is beneficent on the human oral microflora and cytokine level/expression.

ELIGIBILITY:
Inclusion Criteria:

* persons over than 18 years of age with a maximum age of 45 years,
* written informed consent,
* healthy dentition

Exclusion Criteria:

* smoking,
* infectious disease treated with antibiotic in the last two months,
* xerostomia,
* acute oral lesion,
* allergy (lactose),
* systemic or mental condition which contraindicate the participation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-03-16 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Caries preventive action of sour cherry chewing gum | "Through 3 weeks of the study!"
  The action of sour cherry anthocyanins on human salivary microbiome.
Action of sour cherry chewing gum in caries prevention | "During 3 study weeks!"
  The action of sour cherry anthocyanins on cytokine's level.
Effect of sour cherry chewing gum in caries prevention | "Through study completion (3 weeks)!"
  The action of sour cherry anthocyanins on mRNA (messenger ribonucleic acid) expression.

SECONDARY OUTCOMES:
Additional caries preventive action of toothbrush change during sour cherry chewing gum usage | "Till 3 weeks of the study!"
  The effect of toothbrush change on human salivary microbiome.
Additional effect of toothbrush change in caries prevention during sour cherry chewing gum usage | "During 3 study weeks!"
  The effect of toothbrush change on salivary cytokine's level.
Additional action of toothbrush change in caries prevention during sour cherry chewing gum usage | "Through study completion (3 weeks)!"
  The effect of toothbrush change on salivary mRNA expression.

CONTACTS AND LOCATIONS:
Overall Officials: Judit Remenyik, ass. prof., Study Director — University of Debrecen, Institute of Food Technology; Kinga Bágyi, ass. prof., Study Director — University of Debrecen, Faculty of Dentistry
Locations (1):
- University of Debrecen, Debrecen, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Homoki J , Gyemant G , Balogh P , Stundl L , Biro-Molnar P , Paholcsek M , Varadi J , Ferenc F , Kelentey B , Nemes J , Remenyik J . Sour cherry extract inhibits human salivary alpha-amylase and growth of Streptococcus mutans (a pilot clinical study). Food Funct. 2018 Jul 17;9(7):4008-4016. doi: 10.1039/c8fo00064f. PMID 29978173
- [Background] Homoki JR, Nemes A, Fazekas E, Gyemant G, Balogh P, Gal F, Al-Asri J, Mortier J, Wolber G, Babinszky L, Remenyik J. Anthocyanin composition, antioxidant efficiency, and alpha-amylase inhibitor activity of different Hungarian sour cherry varieties (Prunus cerasus L.). Food Chem. 2016 Mar 1;194:222-9. doi: 10.1016/j.foodchem.2015.07.130. Epub 2015 Jul 29. PMID 26471548

DOCUMENTS (1):
  • Informed Consent Form (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/11/NCT05406011/ICF_001.pdf